CLINICAL TRIAL: NCT03059732
Title: Factors Associated With High Mortality of Gastric Adenocarcinoma in Thailand Versus Japan
Status: Completed | Type: Observational
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Collaborators: Osaka Medical Center for Cancer and Cardiovascular Diseases (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, MD, Principle investigator, Gastrointestinal Unit, King Chulalongkorn Memorial Hospital
Other Study IDs: 029/59
Record Dates: First submitted 2017-02-11; First posted 2017-02-23 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Risk Factor
Keywords: Gastric cancer; Thailand; Japan
MeSH Terms: conditions — Stomach Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thailand: Thai patients who diagnosed gastric cancer
  Interventions: Other: Treatment
- Japan: Japanese patients who diagnosed gastric cancer
  Interventions: Other: Treatment

INTERVENTIONS:
Other: Treatment — Observe the treatments of gastric cancer in each group

SUMMARY:
The differences in patient's clinicopathological characteristic between high and low prevalence of gastric cancer region should be further examined to elucidate factors that associate with poor survival rate of patients with gastric cancer. Therefore, this study aimed to evaluate characteristics of patients with gastric adenocarcinoma and factors associated with different outcome in Thailand and Japan to find a clue to improve patients' survival in low prevalence country such as Thailand.

This is a retrospective cohort study. It was conducted at King Chulalongkorn Memorial Hospital, Thailand and Osaka Medical Center for Cancer and Cardiovascular Disease, Japan. Eligible cases were selected by using standardized search protocols: formal computer searches of all patients seen at out-patient clinic and/or hospitalized for gastric cancer between 2010 and 2014.Two physicians, who were informed the definition of each variable, individually reviewed chart of patients.

ELIGIBILITY:
Inclusion Criteria:

* all patients seen at out-patient clinic and/or hospitalized for gastric cancer between 2010 and 2014.

Exclusion Criteria:

* Age < 18 years
* Incomplete data
* Miss diagnosis of gastric adenocarcinoma
* Died from other causes (not related to gastric adenocarcinoma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients seen at out-patient clinic and/or hospitalized for gastric cancer between 2010 and 2014 in King Chulalongkorn Memorial Hospital, Thailand and Osaka Medical Center for Cancer and Cardiovascular Disease, Japan.
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Factors that associated with mortality rate in Thailand compared to Japan | 2010-2014

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Patum Wan, Thailand